CLINICAL TRIAL: NCT06520137
Title: Correlation Between Upper Third Molars Extraction and Upper Second Molars Periodontal Disease: a Prospective Clinical Observational Study
Brief Title: Third Molars Extraction and Periodontal Disease
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Senese (Other)
Responsible Party: Principal Investigator, Malpassi Chiara, Doctor, Azienda Ospedaliera Universitaria Senese
Other Study IDs: 26617
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Tooth Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A with PPD ≤ 3 mm
  Interventions: Procedure: Tooth extraction
- Group B with PPD ≥ 4 mm
  Interventions: Procedure: Tooth extraction

INTERVENTIONS:
Procedure: Tooth extraction — Extraction of maxillary third molars

SUMMARY:
The aim of the study is to evaluate the changes in periodontal conditions on the distal aspect of the second maxillary molar after the extraction of the maxillary wisdom tooth. As secondary outcome patient- related and tooth-related factors will be analysed to evaluate their effects on the periodontal varibales during time.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years or older
* Presence of an impacted upper wisdom tooth that need to undergo surgical extraction
* Participants need to be able to sign and understand the informed consent and to follow the study-related procedures.

Exclusion Criteria:

* People that have compromised general health conditions (ASA 3, 4, 5, 6)
* Patients that assumed antibiotics in the last 6 months
* Pregnant or breastfeeding women
* Patients who suffer from periodontitis stage III and IV
* Presence of a third molar with incomplete root formation is not taken into account for the surgical extraction.
* Smoker patients

Ages: 19 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Hospital population.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Probing Pockeet Depth (PPD) | Baseline, 1 month, 6 months, 12 months, 24 months
  Distance between the free gingival margin and the apical location of the probe's tip.
Bone Level (BL) | Baseline, 1 month, 6 months, 12 months, 24 months
  Distance between the bone crest and the cemento-enamel junction (CEJ)

SECONDARY OUTCOMES:
Type of impaction | Baseline
  According to Archer's classification it is possible to have seven types of impaction: mesio-angular, disto-angular, bucco-angular, linguo-angular, horizontal, vertical, inverted.
Clinical Attachment Level (CAL) | Baseline, 1 month, 6 months, 12 months, 24 months
  Distance between the cemento-enamel junction and the apical location of the probe's tip
Recession (REC) | Baseline, 1 month, 6 months, 12 months, 24 months
  Distance between the free gingival margine and the cemento-enamel junction (CEJ)
Keratinized Tissue (KT) | Baseline, 1 month, 6 months, 12 months, 24 months
  Distance between the muco-gingival line and the free gingival margin

CONTACTS AND LOCATIONS:
Locations (1):
- University of Siena, Siena, Italy/SI, Italy

IPD SHARING:
Plan to Share IPD: Undecided